CLINICAL TRIAL: NCT03386253
Title: Effect of a Non-Invasive Brain Stimulation Technique on Smoking Cessation Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: STUDY00000789
Record Dates: First submitted 2017-11-22; First posted 2017-12-29 (Actual); Results first posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2022-05

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- active tDCS (Experimental): Participants receive active tDCS for five consecutive days before attempting to quit smoking
  Interventions: Device: active tDCS
- sham tDCS (Sham Comparator): Participants receive sham tDCS for five consecutive days before attempting to quit smoking
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: active tDCS — two 13 minute tDCS sessions separated by 20 minutes in between
  Arms: active tDCS
Device: sham tDCS — sham tDCS session given for same length of time as active
  Arms: sham tDCS

SUMMARY:
In this pilot study, the feasibility of using tDCS (a non-invasive brain stimulation technique) while performing a task requiring cognitive flexibility will be examined in smokers and initial data will be collected regarding the effect of tDCS on smoking cessation behaviors. Smokers will be randomized to receive either active or sham tDCS daily for 5 days after which they will attempt to quit smoking. Smoking behavior after the attempted quit date will be assessed at four weekly visits.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 64
* Smoked (on average) at least 5 cigarettes per day
* Be motivated to quit smoking

Exclusion Criteria:

* Unstable medical or psychiatric conditions
* Any medical conditions with neurological sequelae
* History of loss of consciousness of greater than 30 minutes duration or loss of consciousness with neurological sequelae
* Have any medical condition or use any medication that would either increase risk of subjects participating in this study (e.g., medications that lower the seizure threshold) or that would impact measures of interest (e.g. smoking cessation medications).
* Are pregnant or planning to become pregnant during the study
* Current use of pacemaker, intracranial electrodes or implanted defibrillator

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical and Translational Sciences Institute, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 8 | 8
Completed tDCS / Sham Sessions | 7 | 8
Completed (Completed 4 week follow-up session) | 7 | 7
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Number randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (10.3) | 47.0 (13.3) | 45.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Willing to Complete 5 Days of tDCS or Sham
Description: As a feasibility study, the primary endpoint will be to determine if smokers are willing to enroll into and complete a study evaluating tDCS. Number of smokers enrolled and number who complete the 5 day tDCS procedures will be assessed.
Time Frame: 5 days
Population: Number randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
Participants | 7 | 8

2. Secondary Outcome: Change in Number of Cigarettes Smoked Per Day
Description: Change in number of cigarettes smoked per day from the 1 week training period to the 4 week post quit period.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: cigarettes per day
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 7 | 7
cigarettes per day | -4.03 (1.02) | -4.47 (1.09)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; Test type: Superiority; p = 0.77, ANOVA — Group x time p value

ADVERSE EVENTS:
Time Frame: 5 days (time period during which participants received either active or sham tDCS)
Description: Before and after each laboratory session, participants were asked about the presence and severity of 11 specific potential adverse events: 1) Headache; 2) Neck Pain; 3) Scalp Pain; 4) Tingling; 5) Itching; 6) Burning Sensation; 7) Skin Redness; 8) Sleepiness / Fatigue; 9) Poor Concentration; 10) Acute Mood Change; 11) Nausea; 12) An open ended option labeled Other
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/8 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active tDCS (N=8) | Sham tDCS (N=8)
Headache (Nervous system disorders) | 1 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Tingling (Skin and subcutaneous tissue disorders) | 4 | 1
Itching (Skin and subcutaneous tissue disorders) | 2 | 1
Burning sensation (Skin and subcutaneous tissue disorders) | 1 | 2
Sleepiness (General disorders) | 3 | 1
Poor Concentration (Nervous system disorders) | 1 | 3
Mood Change (Psychiatric disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT03386253/Prot_SAP_000.pdf